CLINICAL TRIAL: NCT05775120
Title: Epidemiology of Helicobacter Pylori Infection in Moscow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Other Study IDs: 4/2022-2
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Gastric Atrophy; Gastric Cancer; Helicobacter Pylori Infection
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — gastric mucosa biopsy for OLGA-assessment and culture (H.p. atimicrobal susceptibility)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Screening for H. pylori infection is planned in 5121 citizens living in different administrative districts of Moscow. The cohort will be formed based on age and sex structure of the Moscow population. The presence of H. pylori will be analyzed using 2 non-invasive methods - 13C-urease breath test and serological test (detection of IgG antibodies to H. pylori). An epidemiological questionnaire will be filled out for each respondent which will display basic information on the patient (gender, age, eating habits, bad habits, family history of cancer, etc.), as well as characterize the main symptoms, if any.
  Based on pepsinogen (PG) I levels and PG II (serological markers of atrophy of the gastric mucosa), patients with a high risk of atrophic gastritis and precancerous lesions in the gastric mucosa will be identified and the age and sex structure of atrophic gastritis prevalence in Moscow will be constructed.
- Cohort 2: From 5121 respondents, 500 patients with confirmed H. pylori infection and serological markers of atrophic gastritis and a control group of infected with H. pylori without serological markers of gastric mucosa atrophy will be selected. They will undergo esophagogastroduodenoscopy with two gastric mucosa biopsies. The first will be conducted according to the OLGA system with a pathology assessment of the stage and degree of gastritis, while the second will be taken to determine the antimicrobial susceptibility of H. (polymerase chain reaction and culture). Correlations between serological and patholgy data on atrophy will be assessed in order to determine the reliability of serological screening for atrophy in the Moscow population.
  Interventions: Diagnostic Test: OLGA and H.pylori culture

INTERVENTIONS:
Diagnostic Test: OLGA and H.pylori culture — Upper endoscopy will be performed by endoscopists using modern endoscopes (Fujinon EG-590WR, Olimpus GIF-H190 and others) while patient is sedated. Using sterile biopsy forceps, biopsy specimens will be taken from five areas of the stomach (two biopsy specimens - greater and lesser curvature of the antrum of the stomach; two biopsy specimens - lesser and greater curvature (or anterior and posterior wall) of the body of the stomach and one from the corner of the stomach) for pathology assessment. Pathology assessment of the gastritis stage and degree will be conducted according to the OLGA system developed by the international group of gastroenterologists and pathologists (Atrophy Club).
  Groups: Cohort 2

SUMMARY:
H. pylori is transmitted from individual to individual and causes chronic active gastritis in all infected people. H. pylori infection can result in gastroduodenal ulcers, atrophic gastritis (AG), gastric carcinoma, and gastric MALT lymphoma.

More than 90% of gastric carcinomas are linked to H. pylori infection that causes chronic AG. A long course of the disease leads to the loss of gastric glands (chronic AG) followed by gastric intestinal metaplasia (GIM), dysplasia, and cancer. This defines two cancer prevention strategies: primary that consists of detection and eradication of H. pylori and secondary that focuses on endoscopic screening for pre-neoplastic lesions and follow-up.

Primary prevention planning requires reliable information on the H. pylori prevalence in the population. To design secondary prevention measures, an understanding of the age-sex structure of precancerous changes in the gastric mucosa (the prevalence of atrophic gastritis) is necessary.

H. pylori eradication is the basis of primary prevention of gastric cancer (GC). Approximately 36,000 new cases of GC are registered in the Russian Federation each year, and more than 34,000 patients die from the disease. Men get sick 1.3 times more often than women, the peak incidence occurs at the age of over 50 years. The poor outcomes reflect the late stage of diagnosis of this potentially preventable and treatable cancer. The lack of up-to-date data on the H. pylori prevalence in Moscow hinders developing of measures for the detection and timely treatment of this infection as well as the reduction of GC morbidity and mortality.

DETAILED DESCRIPTION:
Aim: to analyze the prevalence of H. pylori infection and pre-neoplastic lesions in the gastric mucosa in the Moscow population to develop a strategy for gastric cancer and early detection.

Main goals:

1. To determine the prevalence of H. pylori in the Moscow population according to the non-invasive diagnostic method - 13C-urea breath test.
2. To determine the prevalence of H. pylori in the Moscow population according to the serological method - level of IgG antibodies to H.pylori.
3. To assess the prevalence of the gastric mucosa atrophy using serological markers (pepsinogen-I, pepsinogen-II and Gastrin-17) in the different age groups of the Moscow population.
4. To assess the state of the gastric mucosa according to endoscopic and morphological studies using the OLGA system, and their correlation with serological markers of atrophy (pepsinogen I level less than 30 µg/l and/or pepsinogen I/pepsinogen II ratio less than 3).
5. Develop recommendations for GC prevention and early detection strategy.

The planned study will contain two sample cohorts:

Cohort 1 Screening for H. pylori infection is planned in 5121 citizens living in different administrative districts of Moscow. The cohort will be formed based on age and sex structure of the Moscow population. The presence of H. pylori will be analyzed using 2 non-invasive methods - 13C-urease breath test and serological test (detection of IgG antibodies to H. pylori). An epidemiological questionnaire will be filled out for each respondent which will display basic information on the patient (gender, age, eating habits, bad habits, family history of cancer, etc.), as well as characterize the main symptoms, if any.

Based on pepsinogen (PG) I levels and PG II (serological markers of atrophy of the gastric mucosa), patients with a high risk of atrophic gastritis and precancerous lesions in the gastric mucosa will be identified and the age and sex structure of atrophic gastritis prevalence in Moscow will be constructed.

Cohort 2 From 5121 respondents, 500 patients with confirmed H. pylori infection and serological markers of atrophic gastritis and a control group of infected with H. pylori without serological markers of gastric mucosa atrophy will be selected. They will undergo esophagogastroduodenoscopy with two gastric mucosa biopsies. The first will be conducted according to the OLGA system with a pathology assessment of the stage and degree of gastritis, while the second will be taken to determine the antimicrobial susceptibility of H. (polymerase chain reaction and culture). Correlations between serological and patholgy data on atrophy will be assessed in order to determine the reliability of serological screening for atrophy in the Moscow population.

Research methods Diagnostics of H. pylori will be carried out using a modern, non-invasive and accurate method - 13C-urea breath test (13C-UBT).

13C-UBT is recognized as the "gold standard" in the non-invasive diagnosis of H. pylori infection, has a high sensitivity and specificity, above 95%. The test is easy to perform, convenient for patients, and has no side effects.

The main reagent in this test is a solution of urea labeled with the carbon isotope C13. The test is based on the hydrolysis of urea by urease produced by H. pylori that forms ammonia and CO2. After an individual takes a test solution with 13C-labeled urea, 13C-labeled urea, and then 13C carbon dioxide, are absorbed into the bloodstream, enter the lungs and are excreted with exhaled air. Initially, before taking the test solution, the patient's exhaled air is collected in a special sealed bag No. 1. The patient then drinks the test solution. After 30 minutes, a second air sample is exhaled into bag No. 2 that is also hermetically sealed. Then the air samples are analyzed on an infrared spectrometer IR-force 200 that determines the isotope ratio 13С/12С. The increase in labeled CO2 is expressed as delta over baseline (DOB). A DOB greater than 2.0‰ is used as a diagnostic criterion for H. pylori infection.

The infrared (IR) spectrometers of IR-force generation consist of 13C and 12C isotope high selectivity detectors. The specific absorption of CO2 in infrared light with a wavelength of 2-8 microns is used. The spectrometer uses specific optical and mathematical principles to reduce the mutual influence of 13CO2 and 12CO2, which increases the accuracy of the instrument and guarantees the reliability of the entire system. The IR analyzer determines the excess of the 13C/12C ratio over the baseline, i.e. level before taking 13C-urea. In addition, a thermostat is used to maintain a constant temperature and exclude the influence of the external environment.

This test will be conducted in Moscow Clinical Research Center named after A.S. Loginov that is equipped with an IR-force infrared spectrometer and trained specialists.

The second diagnostic test for the presence of H. pylori infection is a serological method - the detection of IgG antibodies to H. pylori. This method is recommended for epidemiological studies but is inferior to the 13C-urease breath test in terms of sensitivity, which is 76% to 84% while the specificity of the method is quite high - 90%. The serological method is based on the detection of specific circulating antibodies to H. pylori in the blood with enzyme immunoassay. The serological analysis will be carried out in Moscow Clinical Research Center named after A.S. Loginov.

Pepsinogens analyses will allow identifying chronic atrophic gastritis and can be used in large-cohorts screening to identify groups of individuals with a high risk of GC, which would require further follow-up with basic endoscopy and pathology investigations. The analysis of PG I provides information on the state of the glands in gastric fundus, PG II - of all parts of the stomach, and their ratio (PG I / PG II) reflects the functional status of the gastric mucosa and closely correlates with the progression of atrophic changes in the gastric mucosa. Normal test results indicate a good condition of the mucous membrane; PG I - 30-165 µg/l, Pepsinogen II - 4 to 22 µg/l, PG I / PG II ratio > 3. Patients with a low concentration of pepsinogen I (<30 ng/ml) and a low PG I / PG II ratio (<3) are likely to have atrophic gastritis of the body of the stomach, precancerous lesions (metaplasia, diplasia), as well as adenocarcinoma that will have to be confirmed by endoscopic and pathology examination. One of the diagnostic sets that assess the serum levels of PG I, PG II, and their ratio (PG I / PG II), as well as determine the concentration of gastrin-17 and the presence of IgG antibodies to H. pylori, is "GastroPanel". The analysis will be carried out in one of the labs of Moscow Clinical Research Center named after A.S. Loginov using enzyme immunoassay.

Upper endoscopy will be performed by endoscopists using modern endoscopes (Fujinon EG-590WR, Olimpus GIF-H190 and others) while patient is sedated. Using sterile biopsy forceps, biopsy specimens will be taken from five areas of the stomach (two biopsy specimens - greater and lesser curvature of the antrum of the stomach; two biopsy specimens - lesser and greater curvature (or anterior and posterior wall) of the body of the stomach and one from the corner of the stomach) for pathology assessment. Pathology assessment of the gastritis stage and degree will be conducted according to the OLGA system developed by the international group of gastroenterologists and pathologists (Atrophy Club).

The stage of atrophy will be assessed on a 4-point scale from 0 to 3, depending on the percentage of atrophied glands. No atrophy (0%) - 0 points, mild atrophy (1-30%) - 1 point, moderate atrophy (31-60%) - 2 points and 3 points - severe atrophy (more than 60%). The obtained data in points will be compared with the developed tables and determine the stage of gastritis from 0 to IV. The degree of gastritis reflects the severity of inflammation, is assessed in the same biopsy specimens by the lymphoplasmacytic and leukocytic infiltration dense in accordance with the visual analog scale, and is expressed in accordance with its assessment table in gradations from 0 to IV.

Number of respondents: 5121 citizens.

Inclusion Criteria:

* Age 18 to 80 years;
* Signed informed consent form.

Criteria for non-inclusion:

* history of taking antibiotics, bismuth-containing drugs within 30 days before the visit and proton pump inhibitors within 14 days before the visit;
* The presence of clinically significant neurological, cardiovascular, gastrointestinal (total of partial gastrectomy), hepatic, renal, immune and other diseases in medical history;
* Patients with diagnosed cancers of any kind who require specialized treatment and/or are currently undergoing anticancer treatment;
* Psychiatric illnesses, including in the past, which, in the opinion of the investigator, make the patient's participation in the study unacceptable;
* Pregnancy;
* Patients who tend to refuse to participate in the study and comply with doctor's recommendations;
* Inability or unwillingness to give informed consent to participate in the study or to fulfill the requirements of the study;

Criteria for exclusion of patients from the study

1. Refusal of further use of the drug;
2. Deterioration of objective indicators of the patient's condition;

Study design The total duration of participation of each patient in the study will be about 2-6 weeks.

Visit 1 (5121 respondents) - day 0: inclusion in the study, informed consent signing, filling out the questionnaire, conducting a 13C-urease breath test, taking a blood test for Gastropanel.

Visit 2 - 500 respondents with serological signs of atrophy (pepsinogen I < 30 ng/ml and/or PGI/PGII < 3 µg/l) and from the control group (14±7 days): EGDS + biopsy according to OLGA.

Expected results

* Large-scale screening of persons for H. pylori infection will allow estimating the actual prevalence of infection among residents of Moscow, which is necessary for planning measures for the primary prevention of gastric cancer.
* Determination of serological markers of atrophy and their correlation with the data of morphological studies will allow assessing the sex and age structure of pre-neoplastic changes in the gastric mucosa, which is necessary to develop an algorithm for secondary prevention of gastric cancer.
* The results of the study will allow developing a comprehensive program for the prevention and early detection of gastric cancer based on an evidence-based combination of primary and secondary prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 to 80 years;

  * Signed informed consent form.

Exclusion Criteria:

* Criteria for non-inclusion:

  * history of taking antibiotics, bismuth-containing drugs within 30 days before the visit and proton pump inhibitors within 14 days before the visit;
  * The presence of clinically significant neurological, cardiovascular, gastrointestinal (total of partial gastrectomy), hepatic, renal, immune and other diseases in medical history;
  * Patients with diagnosed cancers of any kind who require specialized treatment and/or are currently undergoing anticancer treatment;
  * Psychiatric illnesses, including in the past, which, in the opinion of the investigator, make the patient's participation in the study unacceptable;
  * Pregnancy;
  * Patients who tend to refuse to participate in the study and comply with doctor's recommendations;
  * Inability or unwillingness to give informed consent to participate in the study or to fulfill the requirements of the study;

Criteria for exclusion of patients from the study

1. Refusal of further use of the drug;
2. Deterioration of objective indicators of the patient's condition;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Screening for H. pylori infection is planned in 5121 citizens living in different administrative districts of Moscow.
Sampling Method: Non-Probability Sample
Enrollment: 5121 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence of the gastric mucosa atrophy using serological markers | upon inclusion
  (pepsinogen-I, pepsinogen-II and Gastrin-17)
To assess the state of the gastric mucosa according to endoscopic and morphological studies using the OLGA system, and their correlation with serological markers of atrophy | 3 years
  OLGA assessment of biopsy samples (pepsinogen I level less than 30 µg/l and/or pepsinogen I/pepsinogen II ratio less than 3).

SECONDARY OUTCOMES:
To determine the prevalence of H. pylori in the Moscow population according to the non-invasive diagnostic method - 13C-urea breath test. | 3 years
  percent
To determine the prevalence of H. pylori in the Moscow population according to the serological method - level of IgG antibodies to H.pylori. | 3 years
  percent

OTHER OUTCOMES:
Develop recommendations for GC prevention and early detection strategy. | 3 years
  recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry S. Bordin, MD, PhD, Study Director — A.S. Loginov Moscow Clinical Research Center
Locations (1):
- A.S. Loginov Moscow Clinical Scientific Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Result] Sugano K, Tack J, Kuipers EJ, Graham DY, El-Omar EM, Miura S, Haruma K, Asaka M, Uemura N, Malfertheiner P; faculty members of Kyoto Global Consensus Conference. Kyoto global consensus report on Helicobacter pylori gastritis. Gut. 2015 Sep;64(9):1353-67. doi: 10.1136/gutjnl-2015-309252. Epub 2015 Jul 17. PMID 26187502
- [Result] Liou JM, Malfertheiner P, Lee YC, Sheu BS, Sugano K, Cheng HC, Yeoh KG, Hsu PI, Goh KL, Mahachai V, Gotoda T, Chang WL, Chen MJ, Chiang TH, Chen CC, Wu CY, Leow AH, Wu JY, Wu DC, Hong TC, Lu H, Yamaoka Y, Megraud F, Chan FKL, Sung JJ, Lin JT, Graham DY, Wu MS, El-Omar EM; Asian Pacific Alliance on Helicobacter and Microbiota (APAHAM). Screening and eradication of Helicobacter pylori for gastric cancer prevention: the Taipei global consensus. Gut. 2020 Dec;69(12):2093-2112. doi: 10.1136/gutjnl-2020-322368. Epub 2020 Oct 1. PMID 33004546
- [Result] Best LM, Takwoingi Y, Siddique S, Selladurai A, Gandhi A, Low B, Yaghoobi M, Gurusamy KS. Non-invasive diagnostic tests for Helicobacter pylori infection. Cochrane Database Syst Rev. 2018 Mar 15;3(3):CD012080. doi: 10.1002/14651858.CD012080.pub2. PMID 29543326
- [Result] Pimentel-Nunes P, Libanio D, Marcos-Pinto R, Areia M, Leja M, Esposito G, Garrido M, Kikuste I, Megraud F, Matysiak-Budnik T, Annibale B, Dumonceau JM, Barros R, Flejou JF, Carneiro F, van Hooft JE, Kuipers EJ, Dinis-Ribeiro M. Management of epithelial precancerous conditions and lesions in the stomach (MAPS II): European Society of Gastrointestinal Endoscopy (ESGE), European Helicobacter and Microbiota Study Group (EHMSG), European Society of Pathology (ESP), and Sociedade Portuguesa de Endoscopia Digestiva (SPED) guideline update 2019. Endoscopy. 2019 Apr;51(4):365-388. doi: 10.1055/a-0859-1883. Epub 2019 Mar 6. PMID 30841008
- [Result] De Re V, Orzes E, Canzonieri V, Maiero S, Fornasarig M, Alessandrini L, Cervo S, Steffan A, Zanette G, Mazzon C, De Paoli P, Cannizzaro R. Pepsinogens to Distinguish Patients With Gastric Intestinal Metaplasia and Helicobacter pylori Infection Among Populations at Risk for Gastric Cancer. Clin Transl Gastroenterol. 2016 Jul 21;7(7):e183. doi: 10.1038/ctg.2016.42. PMID 27441820
- [Result] Ogutmen Koc D, Bektas S. Serum pepsinogen levels and OLGA/OLGIM staging in the assessment of atrophic gastritis types. Postgrad Med J. 2022 Jun;98(1160):441-445. doi: 10.1136/postgradmedj-2020-139183. Epub 2020 Dec 30. PMID 33380437
- [Result] Megraud F, Bruyndonckx R, Coenen S, Wittkop L, Huang TD, Hoebeke M, Benejat L, Lehours P, Goossens H, Glupczynski Y; European Helicobacter pylori Antimicrobial Susceptibility Testing Working Group. Helicobacter pylori resistance to antibiotics in Europe in 2018 and its relationship to antibiotic consumption in the community. Gut. 2021 Oct;70(10):1815-1822. doi: 10.1136/gutjnl-2021-324032. Epub 2021 Apr 9. PMID 33837118
- [Result] Savoldi A, Carrara E, Graham DY, Conti M, Tacconelli E. Prevalence of Antibiotic Resistance in Helicobacter pylori: A Systematic Review and Meta-analysis in World Health Organization Regions. Gastroenterology. 2018 Nov;155(5):1372-1382.e17. doi: 10.1053/j.gastro.2018.07.007. Epub 2018 Jul 7. PMID 29990487
- [Result] Yue H, Shan L, Bin L. The significance of OLGA and OLGIM staging systems in the risk assessment of gastric cancer: a systematic review and meta-analysis. Gastric Cancer. 2018 Jul;21(4):579-587. doi: 10.1007/s10120-018-0812-3. Epub 2018 Feb 19. PMID 29460004
- [Result] Rugge M, Fassan M, Pizzi M, Zorzetto V, Maddalo G, Realdon S, De Bernard M, Betterle C, Cappellesso R, Pennelli G, de Boni M, Farinati F. Autoimmune gastritis: histology phenotype and OLGA staging. Aliment Pharmacol Ther. 2012 Jun;35(12):1460-6. doi: 10.1111/j.1365-2036.2012.05101.x. Epub 2012 Apr 22. PMID 22519568
- [Result] Sawaki K, Kanda M, Kodera Y. Review of recent efforts to discover biomarkers for early detection, monitoring, prognosis, and prediction of treatment responses of patients with gastric cancer. Expert Rev Gastroenterol Hepatol. 2018 Jul;12(7):657-670. doi: 10.1080/17474124.2018.1489233. Epub 2018 Jun 25. PMID 29902383